CLINICAL TRIAL: NCT00434434
Title: A Phase II, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lyophilized and Aged Liquid Omalizumab in the Prevention of Allergen-Induced Airway Obstruction in Adults With Mild Allergic Asthma
Brief Title: A Study of Omalizumab in the Prevention of Allergen Induced Airway Obstruction in Adults With Mild Allergic Asthma
Acronym: AQUA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q4160g
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Results first posted 2010-05-26 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Allergic Asthma
Keywords: AQUA; anti-CD11; CD11a; Asthma; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: omalizumab
- 2 (Experimental)
  Interventions: Drug: omalizumab
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omalizumab — Aged Liquid; subcutaneous repeating dose
  Arms: 1
Drug: omalizumab — Lyophilized; subcutaneous repeating dose
  Arms: 2
Drug: placebo — Subcutaneous repeating dose
  Arms: 3

SUMMARY:
This was a multicenter, randomized, double-blind, parallel-group, three-arm, placebo-controlled study designed to demonstrate the efficacy of two different formulations of omalizumab compared with placebo in reducing the airway reaction to an inhaled aeroallergen solution in adult subjects with mild allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Meet criteria for the diagnosis of allergic asthma
* Be between the ages of 18 to 65 years
* Have a normal chest X-ray within 2 years of screening

Exclusion Criteria:

* Need daily controller medication for asthma
* History of hypersensitivity to the study drug or to drugs with similar chemical structures or to any ingredients, including excipients of the study medication or drugs related to omalizumab (e.g., monoclonal antibodies, polyclonal gamma globulin)
* Have a documented medical history of anaphylaxis
* Have lung disease other than mild allergic asthma
* Have taken other investigational drugs within 30 days or 5 half-lives prior to the screening visit, whichever is longer
* Are unable or unwilling to comply with study procedures and visits
* Are pregnant or lactating
* Have significant medical illness other than asthma, including malignancies, parasitic infections, immune system disorders, and thrombocytopenia
* Have been treated with omalizumab within 12 months prior to screening
* Currently smoke or have a history of smoking more than 10 pack-years
* Have a history of drug or alcohol abuse, which, in the judgment of the investigator, may put the subject at risk for being unable to participate fully in the study for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wong, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Liquid Omalizumab: Liquid omalizumab subcutaneously either every 2 weeks or every 4 weeks based on their weight and IgE levels at screening
- Lyopholized Omalizumab: Lyophilized omalizumab subcutaneously either every 2 weeks or every 4 weeks based on their weight and IgE levels at screening
- Placebo: Lyophilized placebo subcutaneously either every 2 weeks or every 4 weeks based on their weight and IgE levels at screening
Period: Overall Study
Arm/Group | Liquid Omalizumab | Lyopholized Omalizumab | Placebo
Started | 23 | 24 | 14
Completed | 21 | 24 | 13
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid Omalizumab | Lyopholized Omalizumab | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 14 | 61
Age, Customized [Number; unit: participants]
  18 to 40 years | 18 | 21 | 11 | 50
  41 to 65 years | 5 | 1 | 3 | 9
  > 65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (10.3) | 30.6 (12.8) | 32.0 (9.6) | 30.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 10 | 28
  Male | 13 | 16 | 4 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Logarithmically Transformed (log2) Allergen PC15 Concentration (Allergen Concentration Required to Evoke a 15% Decrease in FEV1)
Description: The primary analysis included two tests: a test for superiority of the lyophilized formulation of omalizumab compared with placebo in the change of allergen concentration and a test for the superiority of the aged liquid omalizumab compared with placebo. The difference for the change in the allergen concentration between the lyophilized formulation of omalizumab and placebo, and between the aged liquid omalizumab and placebo were assessed by the exact Wilcoxon-Mann-Whitney test.
Time Frame: From baseline to Week 16
Population: Modified intent-to-treat (ITT) population
Measure: Median (Full Range); unit: concentration change
Arm/Group | Liquid Omalizumab | Lyopholized Omalizumab | Placebo
Number analyzed (Participants) | 22 | 23 | 13
concentration change | 1.15 [-2.30 to 4.03] | 1.85 [-1.10 to 3.50] | 0.36 [-1.09 to 3.09]
Statistical Analysis 1: Comparison: Liquid Omalizumab vs Placebo; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney); exact Wilcoxon-Mann-Whitney
Statistical Analysis 2: Comparison: Lyopholized Omalizumab vs Placebo; Test type: Superiority or Other; p = 0.0133, Wilcoxon (Mann-Whitney); exact Wilcoxon-Mann-Whitney

2. Secondary Outcome: Ratio of the Allergen Forced Expiratory Volume at One Second (FEV1) Two-point Slope at the Week 16 Allergen Challenge to the Allergen FEV1 Two-point Slope at the Baseline Allergen Challenge
Description: FEV1 is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity, measured in liters. The allergen FEV1 two-point slope is defined as the final percent change in FEV1 from pre-challenge value divided by the final value of allergen concentration used in the challenge.
Time Frame: From baseline to Week 16
Population: Modified ITT population
Measure: Median (Full Range); unit: ratio of FEV1
Arm/Group | Liquid Omalizumab | Lyopholized Omalizumab | Placebo
Number analyzed (Participants) | 22 | 23 | 13
ratio of FEV1 | 0.52 [-0.09 to 3.18] | 0.29 [-0.26 to 2.08] | 0.95 [0.12 to 2.20]
Statistical Analysis 1: Comparison: Liquid Omalizumab vs Placebo; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney); exact Wilcoxon-Mann-Whitney
Statistical Analysis 2: Comparison: Lyopholized Omalizumab vs Placebo; Test type: Superiority or Other; p = 0.0028, Wilcoxon (Mann-Whitney); exact Wilcoxon-Mann-Whitney

ADVERSE EVENTS:
Description: Safety evaluable population
Arm/Group | Liquid Omalizumab | Lyopholized Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 2/24 | 0/14
Other Adverse Events (participants affected / at risk) | 7/23 | 6/24 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid Omalizumab (N=23) | Lyopholized Omalizumab (N=24) | Placebo (N=14)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid Omalizumab (N=23) | Lyopholized Omalizumab (N=24) | Placebo (N=14)
Chest Discomfort (General disorders) | 0 | 1 | 1
Facial Pain (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 2
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 0
Sinus Headache (Nervous system disorders) | 0 | 0 | 1
Middle Insomnia (Psychiatric disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.